CLINICAL TRIAL: NCT06936111
Title: Effect of Residual Lipid and Inflammation Risk on Atherosclerotic Plaque Progression Under Intensive Lipid-lowering Therapy in Coronary Heart Disease
Brief Title: REsiduAL rISk Under Intensive Lipid-lowering Therapy In Coronary Heart Disease
Acronym: REALISTIC
Status: Recruiting | Type: Observational
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Principal Investigator, Chunfeng Dai, M.D., Shanghai Zhongshan Hospital
Other Study IDs: B2024-377R
Record Dates: First submitted 2025-04-12; First posted 2025-04-20 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Coronary Heart Disease (CHD)
MeSH Terms: conditions — Coronary Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- CHD patients undergoing target lesion PCI: This study will enroll patients with CAD undergoing target lesion PCI, with appropriate non-target lesions near the target lesion, which served as the observed lesions
  Interventions: Diagnostic Test: Assessment of residual cholesterol and inflammatory risk factors

INTERVENTIONS:
Diagnostic Test: Assessment of residual cholesterol and inflammatory risk factors — The prespecifed risk factors include CRP, SAA, TNF-α, IL-6, MCP-1, Lp-PLA2, PCSK-9, Lp(a)

SUMMARY:
Intensive lipid-lowering therapy is a cornerstone treatment for coronary heart disease (CHD). However, coronary plaque progression persists in a subset of patients even under intensive lipid-lowering therapy, which may be associated with residual lipid and inflammatory risks. Current research in this area remains largely confined to post hoc analyses of randomized controlled trials , with a notable scarcity of prospective follow-up cohorts. The investigators propose that establishing a prospective cohort will provide more authentic insights into the associations between residual risk factors and plaque progression. In this project, the investigators aim to establish a well-characterized CHD cohort with comprehensive data collection, good compliance, and an appropriate sample size. By focusing on non-target lesions within the target vessel and utilizing intravascular ultrasound (IVUS), the investigators will investigate the impact of residual lipid and inflammatory risks on plaque progression during intensive lipid-lowering therapy.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with CAD and PCI was successfully performed.
* Presence of non-target lesions near the target lesion (more than 5mm proximal or distal), with stenosis of 20% to 50% and identifiable anatomical markers (e.g., branches, calcifications, stent edges).
* 18 to 75 years old.
* Written informed consent.

Exclusion Criteria:

* Known autoimmune diseases, or taking immunosuppressive drugs for a long time before onset.
* Known familial hypercholesterolemia.
* Critical conditions (e.g., cardiogenic shock, acute heart failure).
* Severe renal insufficiency (eGFR < 30 mL /(min·1.73m2)), or severe hepatic insufficiency (ALT or AST≥3 times the upper limit of normal).
* Severe underlying diseases (such as end-stage malignancies), life expectancy < 1 year.
* Allergic to lipid-lowering medications.
* Pregnant, or trying to become pregnant, and breastfeeding women.
* Other conditions deemed unsuitable for inclusion by the researcher.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will enroll patients with CAD undergoing target lesion PCI, with appropriate non-target lesions near the target lesion, which served as the observed lesions
Sampling Method: Non-Probability Sample
Enrollment: 900 (Estimated)
Dates: Start 2025-07-01 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
coronary plaque progression | 9 to 12 months after PCI
  percent change in plaque volume measured by IVUS

SECONDARY OUTCOMES:
carotid plaque progression | 9 to 12 months after PCI
  measured by carotid ultrasound

OTHER OUTCOMES:
MACE | 9 to 12 months after PCI
  major adverse cardiovascular events

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Zhongshan Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: No
The research involves some confidential content